CLINICAL TRIAL: NCT01738542
Title: CLAU Test Results (CLinical Assessment And Endothelin fUnction Assessment After Endothelin Receptor Antagonist) : Randomized Controlled Clinical Trial of Bosentan for Intermittent Claudication in Peripheral Arterial Disease
Brief Title: Safety and Efficacy Study of Bosentan for Intermittent Claudication in Peripheral Arterial Disease
Acronym: CLAU
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospital Universitario Getafe (Other)
Responsible Party: Principal Investigator, Joaquin de Haro, M.D., Randomized controlled clinical trial of Bosentan in Intermittent Claudication in Peripheral Arterial Disease, Hospital Universitario Getafe
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: NTC25102012; E.C.13/2009.CEIC10 (Other Grant/Funding Number: E.C.13/2009.CEIC10)
Record Dates: First submitted 2012-10-30; First posted 2012-11-30 (Estimated); Last update posted 2012-11-30 (Estimated); Status verified 2012-11

CONDITIONS: Peripheral Arterial Disease
Keywords: Bosentan; Peripheral Arterial Disease
MeSH Terms: conditions — Peripheral Arterial Disease | interventions — Bosentan; Hydroxymethylglutaryl-CoA Reductase Inhibitors

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Antiaggregants & Statins & Antihypertensives & Bosentan (Experimental): Bosentan 62.5 mg/12 hours (first four weeks) and 125 mg/12 hours (eight weeks) plus Antiaggregant therapy (AAS 100mg/d or Clopidogrel 75mg/d), Statins and Antihypertensive therapy
  Interventions: Drug: Bosentan; Drug: Antiaggregant therapy; Drug: Statins; Drug: Antihypertensive therapy
- Antiaggregants & Statins & Antihypertensives (Active Comparator): Antiaggregant therapy (AAS 100 mg/d or Clopidogrel 75 mg/d), Statins, Antihypertensive therapy
  Interventions: Drug: Antiaggregant therapy; Drug: Statins; Drug: Antihypertensive therapy

INTERVENTIONS:
Drug: Bosentan — Bosentan 62.5 mg/12 hours (first four weeks) and 125 mg/12 hours (eight weeks)
  Other Names: Tracleer
  Arms: Antiaggregants & Statins & Antihypertensives & Bosentan
Drug: Antiaggregant therapy — AAS 100mg/d or Clopidogrel 75mg/d
Drug: Statins
Drug: Antihypertensive therapy

SUMMARY:
A prospective study, proof-of concept, randomized, controlled, parallel groups, simple blind was performed in 30 male patients (50-60 years old) with Intermittent Claudication (Rutherford category 1-2) recently diagnosed and clinical manifestations not exceeding 6 months with hypertension and/or dyslipidemia as unique co-morbility disorders. After a period of stabilization of the claudication distance in the Stress test (12.5%, 3.2 km/h) during 2 weeks, were randomized 1:1 to the experimental arm (Bosentan 62.5 mg twice daily/four weeks and 125 mg twice daily/eight weeks) or control group.

ELIGIBILITY:
Inclusion Criteria:

* Arterial hypertension and hypercholesterolemia
* ABI <0,9
* Positive claudiometry with a claudication distance between 50 and 500

Exclusion Criteria:

* surgical patient
* Previous revascularization procedure in the Member studied
* Smoker
* Uncontrolled hypertension
* Cardiac Stress Test unfinished
* Prior DVT
* Concomitant severe disease
* Obesity

Ages: 50 Years to 60 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2009-04; Primary Completion 2010-11 (Actual); Study Completion 2010-11 (Actual)

PRIMARY OUTCOMES:
Change in Absolute Claudication Distance (ACD) respect baseline values | 1 Year
  To determine the efficacy of bosentan on the improvement in the absolute claudication distance in the exercise in patients with Intermittent Claudication due Peripheral Arterial Disease.
  ACD and percentage of change, both for the treatment group and control group, at each visit after baseline : 1 month, 3 months, 6 months and 12 months
Change in flow-mediated arterial dilation (FMAD) respect baseline values | 1 Year
  To determine the efficacy of bosentan on the improvement in the overall endothelin function in patients with Intermittent Claudication due Peripheral Arterial Disease
  FMAD for the treatment group and control group, at each visit after baseline : 1 month, 3 months, 6 months and 12 months

SECONDARY OUTCOMES:
Changes in Analytical plasma values at each visit respect baseline values | 1 Year
  Safety of Bosentan in patients with Intermittent Claudication due Peripheral Arterial Disease.
  Analytical values : plasma electrolyte values, hepatic function, renal function, coagulation profiles, peripheral blood cell count
Change in the ankle brachial index (ABI) respect baseline values | 1 Year
  Efficacy of bosentan on the improvement in the hemodynamic states in patients with Intermittent Claudication due Peripheral Arterial Disease.
  ABI for the treatment group and control group, at each visit after baseline : 1 month, 3 months, 6 months and 12 months
Change in subjective claudication distance (SCD) reported by the patient, as is defined in the Walking Impairment Questionnaire (WIQ), respect baseline values | 1 Year
  Efficacy of bosentan on the improvement of functional status (symptoms of claudication) in patients with Intermittent Claudication due Peripheral Arterial Disease
  SCD for the treatment group and control group, at each visit after baseline : 1 month, 3 months, 6 months and 12 months
Occurrence of Adverse events during the study | 1 Year
  Safety of Bosentan in patients with Intermittent Claudication due Peripheral Arterial Disease.

OTHER OUTCOMES:
Change in the serum levels of Endothelin (ET) respect baseline values | 1 Year
  To determine the efficacy of bosentan on the improvement in the endothelin function in patients with Intermittent Claudication due Peripheral Arterial Disease
Change in the serum levels of C-reactive protein (CRP) respect baseline values | 1 Year
  To determine the efficacy of bosentan on the improvement in inflammatory status in patients with Intermittent Claudication due Peripheral Arterial Disease.
  CRP for the treatment group and control group, at each visit after baseline : 1 month, 3 months, 6 months and 12 months

CONTACTS AND LOCATIONS:
Overall Officials: De Haro Joaquin, MD, PhD, Principal Investigator — Hospital Universitario de Getafe
Locations (1):
- Hospital Universitario de Getafe, Getafe, Madrid, Spain

REFERENCES:
- [Derived] De Haro J, Bleda S, Varela C, Esparza L, Acin F; Bosentan Population-Based Randomized Trial for Clinical and Endothelial Function Assessment on Endothelin Antagonist Therapy in Patients With Intermittent Claudication CLAU Investigators. Effect of Bosentan on Claudication Distance and Endothelium-Dependent Vasodilation in Hispanic Patients With Peripheral Arterial Disease. Am J Cardiol. 2016 Jan 15;117(2):295-301. doi: 10.1016/j.amjcard.2015.10.032. Epub 2015 Nov 6. PMID 26651453